CLINICAL TRIAL: NCT06092229
Title: Palpation Versus TACA ("Thyroid-Airline-Cricoid-Airline") Ultrasonography for Identifying the Cricothyroid Membrane in Case of a Laterally Deviated Larynx
Brief Title: Palpation Versus TACA- Ultrasonography for Identifying the Cricothyroid Membrane in Case of a Laterally Deviated Larynx
Acronym: Devtrach2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Seltz Kristensen, Consultant Anaesthetist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Devtrach2
Record Dates: First submitted 2023-10-14; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Airway Management
Keywords: Airway Management, cricothyrotomy
MeSH Terms: interventions — Palpation; Ultrasonography

STUDY DESIGN:
Intervention Model Description: randomised to either "palpation" or "ultrasonography"
  The participants are thus randomised to use either "palpation" or to use "ultrasonography" to DIAGNOSE the position of the cricothyroid membrane
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palpation (Active Comparator): digital palpation used to identify the cricothyroid membrane
  Interventions: Diagnostic Test: Palpation
- Ultrasonography (Experimental): Ultrasonography (TACA approach) used to identify the cricothyroid membrane
  Interventions: Diagnostic Test: Ultrasonography with TACA approach

INTERVENTIONS:
Diagnostic Test: Palpation — identification of the cricothyroid using PALPATION, a procedure used to prepare for front of neck airway access
  Arms: Palpation
Diagnostic Test: Ultrasonography with TACA approach — identification of the cricothyroid membrane, using ULTRASONOGRAPHY with TACA approach , a procedure used to prepare for front of neck airway access
  Arms: Ultrasonography

SUMMARY:
test persons, anaesthesiologists will identify the cricothyroid membrane on a silicone model of the neck with either palpation or ultrasonography.

The ultrasonographic method to be used is the Thyroid-Airline-Cricoid-Airline (TACA) approach.

The larynx-model is deviated to one of the sides to simulate a patient with neck pathology

DETAILED DESCRIPTION:
test persons, anaesthesiologists will identify the cricothyroid membrane on a silicone model of the neck with either palpation or ultrasonography.

The ultrasonographic method to be used is the Thyroid-Airline-Cricoid-Airline (TACA) approach.

The larynx-model is deviated to one of the sides to simulate a patient with neck pathology.

The test persons are randomised to use other palpation or ultrasonography. Al attempts are video-taped

ELIGIBILITY:
Inclusion Criteria: Participants in a course of airway management -

Exclusion Criteria: Exclusion Criteria: unwillingness to participate

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Correct identification of the cricothyroid membrane within a minute | 1 minute
  The fraction of correct identifications of the location of the cricothyroid membrane

SECONDARY OUTCOMES:
Correct identification of the sagittal plane within the airway | 1 minute
  The fraction of identifications that were within the sagittal boundaries of the trachea

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kristensen, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, department of anaesthesia, Copenhagen, Denmark